CLINICAL TRIAL: NCT01858805
Title: Circulating Tumor Cells as a Biomarker for Preoperative Prognostic Staging in Patients With Esophageal Cancer
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. med. Matthias Reeh, MD, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: CTC-EC; 184 (Other Grant/Funding Number: HAMBURGER STIFTUNG ZUR FÖRDERUNG DER KREBSBEKÄMPFUNG)
Record Dates: First submitted 2013-05-14; First posted 2013-05-21 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Resectable Esophageal Cancer
Keywords: esophagus carcinoma; surgery; circulating tumor cells
MeSH Terms: conditions — Esophageal Neoplasms; Neoplastic Cells, Circulating | interventions — Esophagectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- detection of circulating tumors cells: This prospective, single-institution study conducted at the University Hospital Hamburg-Eppendorf (Hamburg, Germany) enrolled 123 patients with ECs that were initially considered resectable. Only patients with histologically proven EC were included. Peripheral blood samples for CTC analysis were collected immediately before surgery.
  Interventions: Procedure: esophagectomy

INTERVENTIONS:
Procedure: esophagectomy

SUMMARY:
Despite the availability of several preoperative diagnostic techniques, accurate pretreatment staging of esophageal cancer (EC) remains challenging. Therefore, The investigators evaluated the prognostic significance of circulating tumor cells (CTCs) in patients with EC.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* resectable esophageal cancer

Exclusion Criteria:

* < 18 years
* esophageal cancer with preoperative distant metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective, single-institution study conducted at the University Hospital Hamburg-Eppendorf (Hamburg, Germany) enrolled 123 patients with ECs that were initially considered resectable.
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2010-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
overall survival | 2 years

SECONDARY OUTCOMES:
recurrence-free survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hamburg-Eppendorf, Hamburg, Germany